CLINICAL TRIAL: NCT01819844
Title: Subcutaneous Continuous Glucose Monitoring and Intravenous Dosing of Insulin and Dextrose for Automated Glycemic Control in the Inpatient Setting
Brief Title: Inpatient Closed-loop Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011P000993
Record Dates: First submitted 2013-02-28; First posted 2013-03-28 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus; Hyperglycemia
Keywords: Closed-loop blood glucose control; Continuous glucose monitoring; Bionic pancreas; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed-loop blood glucose control (Experimental): Type 1 diabetes, Type 2 diabetes, total daily dose (TDD) of insulin that is > 1 u/kg or > 2 u/kg.
  Interventions: Device: Closed-loop blood glucose control

INTERVENTIONS:
Device: Closed-loop blood glucose control — The InPatient Closed Loop Device is made up of the three components; the Abbott FreeStyle Navigator subcutaneous continuous glucose monitor, the Symbiq insulin-dextrose infusion system, and the control algorithm. In this feasibility trial we will study 6 insulin-sensitive subjects with type 1 diabetes and 6 subjects with type 2 diabetes and a high insulin requirement (3 with total daily dose from 1-1.9 u/kg and 3 with total daily dose > 2 u/kg).
  Other Names: InPatient Closed-Loop Blood Glucose Control Device.

SUMMARY:
The purpose of this study is to test an experimental medical device designed to automatically control blood sugar. This device was designed for use by patients with diabetes while they are in the hospital, and others who may develop high blood sugar as a result of their medical problems.

DETAILED DESCRIPTION:
The goal of this first-in-man trial is to test the safety and efficacy of the automated, closed-loop control system in insulin sensitive subjects with type 1 diabetes, insulin sensitive subjects with type 2 diabetes (TTD > 1u/kg/day), and subjects with type 2 diabetes and substantial insulin resistance (<2 u/kg/day). The results of this study will help to design future studies, exploring the use of the closed-loop system for BG control in hospitalized patients, including those with diabetes or hyperglycemia of critical illness.

ELIGIBILITY:
Inclusion Criteria

Subjects with type 1 diabetes

* Age 21 to 75 with clinical type 1 diabetes for at least one year
* Diabetes managed using an insulin infusion pump and rapid- or very-rapid-acting insulins
* Total daily dose (TDD) of insulin that is < 1 u/kg

Subjects with type 2 diabetes

* Age 21 to 75 with clinical type 2 diabetes for at least one year
* Diabetes managed using NPH as the basal insulin, which may be supplemented with regular or rapid-acting insulin
* Total daily dose (TDD) of insulin that is > 1 u/kg/day but < 2 u/kg/day or > 2 u/kg/day

Exclusion Criteria:

* Pregnancy
* Renal insufficiency
* Cancer
* Abnormal EKG suggestive of coronary artery disease or increased risk of malignant arrhythmia
* Acute illness or exacerbation of chronic illness at the time of the study procedure
* Use of non-insulin, injectable anti-diabetic medications or oral anti-diabetic medications other than metformin
* History of allergy or adverse reaction to aspirin, peptic ulcers or bleeding disorders
* Known history of coronary artery disease, TIA or stroke
* History of seizures
* Transaminitis
* Stage 2 hypertension at the time of screening

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Diabetes Research Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.bionicpancreas.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed-loop Blood Glucose Control
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Average Blood Glucose Over the Closed-loop Control Period, as Determined From GlucoScout Measurements.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
mg/dl
  Overall average blood sugar | 115.9 (19.7)
  Type 1 subjects average blood sugar | 107.0 (13.6)
  Type 2 subjects average blood sugar | 124.83 (21.85)

2. Secondary Outcome: Number of Carbohydrate Interventions (15 g) Delivered According to Study Protocol
Time Frame: 12 hours
Measure: Number; unit: number of carbohydrate interventions
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
number of carbohydrate interventions | 0

3. Secondary Outcome: Number of BG Events < 70 mg/dl and Nadir BG for Each as Determined Form GlucoScout Measurements
Time Frame: 12 hours
Measure: Number; unit: Blood glucose values < 70 mg/dl
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
Blood glucose values < 70 mg/dl | 4

4. Secondary Outcome: Fraction of Time Spent Within Each of the Following Glucose Ranges as Determined From GlucoScout Measurements: - < 70 mg/dl - 70-120 mg/dl - 70-180 mg/dl - >180 mg/dl
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
percentage of time
  70-180 mg/dl | 95.5 (7.6)
  70-120 mg/dl | 67.5 (27.7)
  < 70 mg/dl | 0.25 (0.45)
  > 180 mg/dl | 4.3 (7.8)

5. Secondary Outcome: Average Blood Glucose Over the Closed-loop Control Period as Determined From the CGM Driving the Control Algorithm
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
mg/dl | 115.8 (21.4)

6. Secondary Outcome: Number of BG Events < 70 mg/dl as Determined by the CGM
Time Frame: 12 hours
Measure: Number; unit: events
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
events | 8

7. Secondary Outcome: Fraction of Time Spent Within Each of the Following Glucose Ranges as Determined From the CGM Driving the Control Algorithm: o < 70 mg/dl o 70-120 mg/dl o 70-180 mg/dl o >180 mg/dl
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
percentage of time
  < 70 mg/dl | 1.5 (3.0)
  70-120 mg/dl | 66.8 (26.4)
  70-180 mg/dl | 94.4 (6.9)
  > 180 mg/dl | 4.0 (7.3)

8. Secondary Outcome: Insulin Dosing (u/kg)
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: units/kilogram
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
units/kilogram | 0.42 (0.28)

9. Secondary Outcome: Dextrose Dosing (g/kg)
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: grams/kilogram
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
grams/kilogram | 0.48 (0.45)

10. Secondary Outcome: Accuracy of the CGM Device Using the GlucoScout Measurements as the Standard.
Description: The Mean Absolute Relative Difference (MARD) between CGM and Glucoscout
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: percent absolute relative difference
Arm/Group | Closed-loop Blood Glucose Control
Number analyzed (Participants) | 12
percent absolute relative difference | 8.29 (7.41)

ADVERSE EVENTS:
Arm/Group | Closed-loop Blood Glucose Control
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No